CLINICAL TRIAL: NCT03759834
Title: Cochlear Promontory Stimulation for Treatment of Tinnitus: Towards Developing an Implantable Device
Brief Title: Cochlear Promontory Stimulation for Treatment of Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Matthew L. Carlson, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-004832; PR180961 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2017-11-30; First posted 2018-11-30 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Masking Description: The electrode will be placed in the middle ear. The patient and investigator will be blinded to the "on-off" status of the device. The patient will report if they have improvement of their tinnitus while both the patient and investigator are blinded to the "on-off" status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Testing Arm (Experimental): There will only be one arm. The patient and investigator will initially be blinded to the "on-off" status of the electrode. The patient will thus serve as an internal control for testing. Once device integrity and possible benefit is confirmed, the patients will undergo non-tactile electrical stimulation to the bone of the inner ear (cochlear promontory) for short term relief of tinnitus via Cochlear promontory stimulation.
  Interventions: Device: Cochlear promontory stimulation

INTERVENTIONS:
Device: Cochlear promontory stimulation — Promontory stimulation is an established otologic procedure that was initially developed as a diagnostic tool to assess patient candidacy for cochlear implantation. Promontory stimulation is most commonly performed in the outpatient setting on an awake patient by placing a single insulated probe through a topically anesthetized tympanic membrane and applying monopolar current for several seconds to minutes. The initial session of promontory stimulation will define optimal stimulation parameters (i.e., location, current level, pulse-width, phase polarity), where maximal tinnitus suppression occurs with minimal or no auditory percept. Additional stimulation testing visits will confirm these findings.

SUMMARY:
Tinnitus is the perception of sound when no external noise is present. The Center for Disease Control (CDC) estimates over 50 million - nearly 15% of the general public -experience some form of tinnitus. Roughly 20 million people struggle with burdensome chronic tinnitus, with 2 million experiencing extreme and debilitating symptoms.

The 2014 Clinical Practice Guideline on tinnitus from the American Academy of Otolaryngology - Head and Neck Surgery summarized the existing state of tinnitus management by stating "A cure for primary tinnitus does not yet exist, and despite claims to the contrary, no method has been proven to provide long-term suppression of tinnitus."

The purpose of this study is to look at the safety and efficacy of cochlear promontory stimulation in the short term relief of tinnitus. The secondary goal of the study is to determine the optimum region(s) of the cochlear promontory in planning for an implantable electrical device for long term tinnitus suppression.

DETAILED DESCRIPTION:
Candidate subjects will undergo a temporal bone Computed Tomography (CT) scan, contrast enhanced head Magnetic Resonance Imaging (MRI), audiogram with immittance testing, pitch and level matching of tinnitus, Distortion Product Otoacoustic Emissions (DPOAE) and Auditory Brainstem Response (ABR) testing prior to promontory stimulation. Head MRI, DPOAE, audiogram and immittance testing are considered clinically routine for assessment of asymmetric tinnitus. Temporal bone CT, ABR, tinnitus pitch, level matching, masking levels and residual inhibition testing are not standard clinical assessments for asymmetric tinnitus. In addition, subjects will complete the Tinnitus Handicap Inventory (THI), Tinnitus Functional Index (TFI) and Visual Analog Scale (VAS) questionnaires three separate times within the week prior to promontory stimulation testing. Additional testing for comorbid anxiety and depressive conditions will be a screening Generalized Anxiety Disorder (GAD7), Patient Health Questionnaire (PHQ8), and short Health Anxiety Inventory (HAI-S). The NEO Personality Inventory (NEO PI) will be administered to provide baseline information. The initial session of promontory stimulation will define optimal stimulation parameters (i.e., location, current level, pulse-width, phase polarity), where maximal tinnitus suppression occurs with minimal or no auditory percept. After these parameters are established, the patient will complete the THI, TFI, and VAS immediately prior to stimulation, during stimulation, and following completion of stimulation at 10-minutes, 1-hour, 24-hours, 48-hours, and 1-week following completion of stimulation. In addition, pitch and level matching of tinnitus will be completed immediately upon completion of each promontory stimulation session. Each patient will undergo three successive treatments separated by 1-week. Prior to each treatment, the patient will receive an audiogram and DPOAE testing to document interval safety. At the conclusion of the study, subjects will be asked about their willingness to undergo surgical implantation of a device capable of long-term scheduled or on-demand electrical stimulation for tinnitus suppression

ELIGIBILITY:
Inclusion Criteria:

1. Normal to moderate sensorineural hearing loss (based on pure tone audiometry (PTA) of 500, 1000 and 2000 Hz) and a word recognition score equal to or greater than 60%
2. Asymmetric or unilateral subjective tonal tinnitus
3. Tinnitus that is disruptive

   1. Determined by THI score (in the severe range i.e. ≥56/100)
   2. TFI (in the severe range i.e. ≥52/100)
   3. Tinnitus VAS (≥ 5/10 )
4. Tinnitus that is intractable, and has not been ameliorated by conventional measures such as a hearing aid or masking
5. Normal contrast-enhanced MRI of the head

Exclusion Criteria:

1. Tinnitus present less than 6 months or longer than 12 years; it is permissible to include people who have had intermittent or constant tinnitus longer than 12 years as long as it was not perceived as severe longer than 12 years
2. History of brain or major ear surgery
3. Prior major head trauma
4. Ongoing clinical diagnosis of depression or anxiety; for the purposes of this study, it is permissible to include people who: 1. have a past history of clinically diagnosed depression or anxiety that is no longer currently active; or 2. people who have depressive or anxious symptoms that are thought to primarily result from severe tinnitus

   a. Determined by screening using the GAD 7, PHQ8, and HAI-S
   * GAD7 > 9 (indicates clinically significant anxiety)
   * PHQ > 9 (indicates clinically significant depression)
   * HAI-S > 25 (hypochondriacal level illness anxiety)
5. Inability to assess, continue or complete trial
6. Currently on regularly scheduled antidepressants, anxiolytics or antipsychotics; for this study, it is permissible to include people who use such medications at lower doses as a sleep aid or for people who intermittently use such medications for situational anxiety (e.g., Ativan before airplane travel)
7. Active use of other tinnitus treatments; for the purposes of this study it is permissible to include people who prefer to use a hearing aid to amplify ipsilateral hearing loss
8. Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Carlson, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tunkel DE, Bauer CA, Sun GH, Rosenfeld RM, Chandrasekhar SS, Cunningham ER Jr, Archer SM, Blakley BW, Carter JM, Granieri EC, Henry JA, Hollingsworth D, Khan FA, Mitchell S, Monfared A, Newman CW, Omole FS, Phillips CD, Robinson SK, Taw MB, Tyler RS, Waguespack R, Whamond EJ. Clinical practice guideline: tinnitus. Otolaryngol Head Neck Surg. 2014 Oct;151(2 Suppl):S1-S40. doi: 10.1177/0194599814545325. PMID 25273878
- [Background] Tsai BS, Sweetow RW, Cheung SW. Audiometric asymmetry and tinnitus laterality. Laryngoscope. 2012 May;122(5):1148-53. doi: 10.1002/lary.23242. Epub 2012 Mar 23. PMID 22447577
- [Background] Perez R, Shaul C, Vardi M, Muhanna N, Kileny PR, Sichel JY. Multiple electrostimulation treatments to the promontory for tinnitus. Otol Neurotol. 2015 Feb;36(2):366-72. doi: 10.1097/MAO.0000000000000309. PMID 24691511
- [Background] Rubinstein JT, Tyler RS, Johnson A, Brown CJ. Electrical suppression of tinnitus with high-rate pulse trains. Otol Neurotol. 2003 May;24(3):478-85. doi: 10.1097/00129492-200305000-00021. PMID 12806303
- [Background] Watanabe K, Okawara D, Baba S, Yagi T. Electrocochleographic analysis of the suppression of tinnitus by electrical promontory stimulation. Audiology. 1997 May-Jun;36(3):147-54. doi: 10.3109/00206099709071968. PMID 9193732
- [Background] Steenerson RL, Cronin GW. Treatment of tinnitus with electrical stimulation. Otolaryngol Head Neck Surg. 1999 Nov;121(5):511-3. doi: 10.1016/S0194-5998(99)70048-3. PMID 10547461
- [Background] Mertens G, De Bodt M, Van de Heyning P. Cochlear implantation as a long-term treatment for ipsilateral incapacitating tinnitus in subjects with unilateral hearing loss up to 10 years. Hear Res. 2016 Jan;331:1-6. doi: 10.1016/j.heares.2015.09.016. Epub 2015 Oct 24. PMID 26433053
- [Background] Tyler RS. Patient preferences and willingness to pay for tinnitus treatments. J Am Acad Audiol. 2012 Feb;23(2):115-25. doi: 10.3766/jaaa.23.2.6. PMID 22353680
- [Background] Arts RA, George EL, Stokroos RJ, Vermeire K. Review: cochlear implants as a treatment of tinnitus in single-sided deafness. Curr Opin Otolaryngol Head Neck Surg. 2012 Oct;20(5):398-403. doi: 10.1097/MOO.0b013e3283577b66. PMID 22931903
- [Background] Arts RA, George EL, Chenault MN, Stokroos RJ. Optimizing intracochlear electrical stimulation to suppress tinnitus. Ear Hear. 2015 Jan;36(1):125-35. doi: 10.1097/AUD.0000000000000090. PMID 25090456
- [Background] Zeman F, Koller M, Figueiredo R, Aazevedo A, Rates M, Coelho C, Kleinjung T, de Ridder D, Langguth B, Landgrebe M. Tinnitus handicap inventory for evaluating treatment effects: which changes are clinically relevant? Otolaryngol Head Neck Surg. 2011 Aug;145(2):282-7. doi: 10.1177/0194599811403882. PMID 21493265
- [Background] Topf MC, Hsu DW, Adams DR, Zhan T, Pelosi S, Willcox TO, McGettigan B, Fisher KW. Rate of tympanic membrane perforation after intratympanic steroid injection. Am J Otolaryngol. 2017 Jan-Feb;38(1):21-25. doi: 10.1016/j.amjoto.2016.09.004. Epub 2016 Sep 28. PMID 27751619
- [Derived] Marinelli JP, Anzalone CL, Prummer CM, Poling GL, Staab JP, Tombers NM, Lohse CM, Carlson ML. Electrical stimulation of the cochlea for treatment of chronic disabling tinnitus: an open-label trial towards the development of an implantable device. J Transl Med. 2022 Jan 29;20(1):56. doi: 10.1186/s12967-022-03271-4. PMID 35093126
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants withdrew consent prior to starting treatment.
Groups:
- Testing Arm: There was one arm. The patient and investigator were initially blinded to the "on-off" status of the electrode. The patient served as an internal control for testing. Once device integrity and possible benefit was confirmed, the patients underwent non-tactile electrical stimulation to the bone of the inner ear (cochlear promontory) for short term relief of tinnitus via Cochlear promontory stimulation.
  Cochlear promontory stimulation: Promontory stimulation is an established otologic procedure that was initially developed as a diagnostic tool to assess patient candidacy for cochlear implantation. Promontory stimulation is most commonly performed in the outpatient setting on an awake patient by placing a single insulated probe through a topically anesthetized tympanic membrane and applying monopolar current for several seconds to minutes. The initial session of promontory stimulation will define optimal stimulation parameters (i.e., location, current level, pulse-width, phase polarity), where maximal tinnitus suppression occurs with minimal or no auditory percept. Additional stimulation testing visits will confirm these findings.
Period: Overall Study
Arm/Group | Testing Arm
Started | 22
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Testing Arm
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Short Term Relief of Tinnitus as Measured by the Tinnitus Handicap Inventory
Description: The Tinnitus Handicap Inventory (THI) has 25 questions with possible answers of Yes (4 points), Sometimes (2 points), and No (0 points). Scores categories are (1-16: Slight or no handicap - Grade 1), (18-36: Mild handicap - Grade 2), (38-56: Moderate handicap - Grade 3), (58-76: Severe handicap - Grade 4), (78-100: Catastrophic handicap - Grade 5). Total score ranges from 0 to 100 with higher scores indicating a worse outcome.
Time Frame: Baseline to 4 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Testing Arm
Number analyzed (Participants) | 22
score on a scale | -31 [-38 to -25]

2. Secondary Outcome: Optimal Location of Tinnitus Relief
Description: Location on the cochlear promontory where highest perceived benefit from electrical stimulation
Time Frame: Immediately after electrical stimulation procedure (approximately 1 min after stimulation)
Population: No participants were measured and analyzed for this outcome measure because the principal investigator decided to only use one standard location on the promontory during the study for all participants.
Arm/Group | Testing Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: Auditory Feedback
Description: The number of subjects that reported hearing the electrical stimulus (if at all)
Time Frame: Immediately after electrical stimulation procedure (approximately 1 min after stimulation)
Measure: Count of Participants; unit: Participants
Arm/Group | Testing Arm
Number analyzed (Participants) | 22
Participants | 22

4. Secondary Outcome: Tactile Feedback
Description: The number of subjects that reported feeling the electrical stimulus (if at all)
Time Frame: Immediately after electrical stimulation procedure (approximately 1 min after stimulation)
Measure: Count of Participants; unit: Participants
Arm/Group | Testing Arm
Number analyzed (Participants) | 22
Participants | 22

5. Secondary Outcome: Change in Short Term Relief of Tinnitus as Measured by the Tinnitus Functional Index
Description: The Tinnitus Functional Index (TFI) contains eight subscales (domains), of which seven contain 3 items and one contains 4. The possible responses for each item range from 0 (did not interfere) to 10 (completely interfered). The total score is transformed to a scale ranging from 0 (no interference) to 100 (completely interfered with activities).
Time Frame: Baseline to 4 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Testing Arm
Number analyzed (Participants) | 22
score on a scale | -35 [-42 to -28]

6. Secondary Outcome: Change in Short Term Relief of Tinnitus as Measured by the Visual Analog Scale
Description: The Visual Analog Scale (VAS) for Numeric Pain Distress was used for this outcome. The VAS is a 11-item questionnaire assessing pain. Using a scale of 0 (no pain) and 10 (unbearable pain). Total scores range from 0 - 110, lower scores indicating lower pain and higher scores indicating greater pain.
Time Frame: Baseline to 4 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Testing Arm
Number analyzed (Participants) | 22
score on a scale | -3.7 [-4.7 to -2.8]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of informed consent through study completion, approximately 4 months.
Arm/Group | Testing Arm
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT03759834/Prot_SAP_001.pdf
  • Informed Consent Form (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT03759834/ICF_000.pdf